CLINICAL TRIAL: NCT07140471
Title: Comparison of Sublay Versus Onlay Mesh Repair for Ventral Abdominal Wall Hernia: A Randomized Controlled Trial
Brief Title: Comparison of Sublay and Onlay Mesh Repair in Ventral Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Ehsan ullah (Other)
Responsible Party: Sponsor-Investigator, Sana Ehsan ullah, Principal Investigator and Senior Registrar, Recep Tayyip Erdogan Hospital Pakistan
Organization: Recep Tayyip Erdogan Hospital Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHHN_IRB_2023_05_026
Record Dates: First submitted 2025-08-06; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ventral Hernia; Incisional Hernia
Keywords: Sublay Mesh Repair; Onlay Mesh Repair; Polypropylene Mesh; Hernia Surgery; Wound Infection; Seroma Formation; Hernia Recurrence; Randomized Controlled Trial; Open Hernia Repair
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia; Wound Infection

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel arms: one receiving onlay mesh repair and the other receiving sublay mesh repair.
Masking Description: This was an open-label study with no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay Mesh Repair (Active Comparator): Participants underwent onlay mesh repair, where the polypropylene mesh was placed over the anterior rectus sheath after hernia reduction and defect closure.
  Interventions: Procedure: Onlay Mesh Repair
- Sublay Mesh Repair (Experimental): Participants underwent sublay mesh repair, where the polypropylene mesh was placed in the retrorectus space after posterior sheath dissection.
  Interventions: Procedure: Sublay Mesh Repair

INTERVENTIONS:
Procedure: Onlay Mesh Repair — Polypropylene mesh is placed over the anterior rectus sheath and fixed with Prolene sutures after hernia sac reduction.
  Arms: Onlay Mesh Repair
Procedure: Sublay Mesh Repair — Polypropylene mesh placed in the retrorectus space and fixed with Prolene sutures after Rectus Sheath Dissection
  Arms: Sublay Mesh Repair

SUMMARY:
This study is designed to compare two different surgical methods for repairing ventral abdominal wall hernias: sublay mesh repair and onlay mesh repair. Ventral hernias are common and occur when tissue pushes through a weak spot in the abdominal wall. Both sublay and onlay techniques involve placing a synthetic mesh to strengthen the abdominal wall, but the position of the mesh differs. This trial will evaluate postoperative outcomes, including surgical wound infections, seroma (fluid buildup), and hernia recurrence, over a six-month follow-up period. The findings are expected to help inform surgical decision-making, particularly in resource-limited hospitals.

DETAILED DESCRIPTION:
This prospective, open-label, randomized controlled trial aims to compare outcomes between sublay and onlay mesh repair techniques in patients with ventral abdominal wall hernias. The study is being conducted at Recep Tayyip Erdogan Hospital, Muzaffargarh, Pakistan, from February 2022 to August 2023. A total of 96 patients aged 18-60 years with primary or incisional ventral hernias (defect size 40-100 mm) are included. Patients are randomized into two groups: Group A undergoes onlay mesh repair, and Group B undergoes sublay mesh repair. Both procedures involve placement of macroporous polypropylene mesh with appropriate overlap and standard fixation techniques.

Primary outcomes include wound infection (as per CDC criteria), seroma formation (confirmed by ultrasound), and hernia recurrence (clinically and via ultrasonography) at six-month follow-up. Secondary outcomes include operative time, postoperative pain (measured via visual analog scale), and hospital stay duration. Data analysis will be performed using SPSS v26.0.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 60 years

Primary or incisional ventral abdominal wall hernia

Hernia defect size between 40-100 mm

Duration of hernia ≥6 months

Suitable for open mesh hernioplasty

Written informed consent provided

Exclusion Criteria:

Diabetes mellitus >5 years

Chronic liver disease

Obstructed or strangulated hernia

Immunocompromised status

Severe cardiopulmonary disease or contraindications to general anesthesia

Pregnant or lactating women

Inability to attend follow-up visits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical wound infection | Within 30 days after surgery
  Wound infection was assessed based on CDC criteria: fever >38°C, erythema, purulent discharge, or swelling at the surgical site. Evaluated daily during hospitalization and at 2-week follow-up.
Incidence of seroma formation | Within 30 days postoperatively
  Seroma defined as subcutaneous fluid accumulation confirmed by clinical exam and ultrasonography. Evaluated during follow-up visits.
Hernia recurrence rate | 6-month follow-up
  Recurrence assessed through physical examination and confirmed via ultrasonography at 6 months after surgery.

SECONDARY OUTCOMES:
Mean operative time | Time in minutes from skin incision to skin closure, recorded intraoperatively.
  During surgery
Length of postoperative hospital stay | From the day of surgery until hospital discharge (average of 3-7 days).
  Number of days from surgery to discharge recorded for each participant.
Postoperative pain score | At 6 hours, 24 hours, and 48 hours after surgery, and then every 48 hours thereafter until hospital discharge
  Pain evaluated using the visual analog scale (VAS) from 0 (no pain) to 10 (worst pain) during inpatient stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan Hospital, Muzaffargarh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to privacy concerns, institutional policy, and the absence of specific data-sharing agreements or infrastructure for secure dissemination.